CLINICAL TRIAL: NCT02802631
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics of Minocin® (Minocycline) for Injection in Healthy Adult Subjects
Brief Title: Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Minocin (Minocycline) for Injection in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rempex (a wholly owned subsidiary of Melinta Therapeutics, Inc.) (Industry)
Collaborators: Universitätsklinikum Köln (Other); Innovative Medicines Initiative (Other)
Responsible Party: Sponsor
Organization: Melinta Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDCO-MIN-16-02; 701 (IMI WP8A ID #) (Other: The Medicines Company)
Record Dates: First submitted 2016-06-09; First posted 2016-06-16 (Estimated); Results first posted 2023-05-09 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Normal Healthy Volunteers
Keywords: Bacterial infections
MeSH Terms: conditions — Bacterial Infections | interventions — Minocycline; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Intervention Model Description: Model Description: Cohorts 1 and 2 were run concurrently as they were using the approved doses of intravenous minocycline in the United States. Cohorts 3, 4, 5 and 6 were run sequentially and only after review of data from the preceding cohorts by the data monitoring committee.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minocin (minocycline) for Injection (Experimental): Minocin (minocycline) for Injection was supplied as a sterile lyophilized powder in single-use 10-milliliter (mL) glass vials. Each vial contained 108 milligrams (mg) of minocycline hydrochloride equivalent to 100 mg of minocycline. Each cohort received one of the following dosages of Minocin (minocycline) for Injection: 100 mg, 200 mg, 300 mg, 400 mg, 500 mg, or 600 mg. Within each cohort, participants received a single dose on Day 1, followed by 7 days of multiple doses (Days 4 to 10, given every 12 hours), followed by a single dose on Day 11.
  Interventions: Drug: Minocin (minocycline) for Injection
- 0.9% Sodium Chloride Injection USP (Placebo Comparator): Placebo was in the form of the same 100-mL bags of normal saline (0.9% Sodium Chloride Injection United States Pharmacopeia [USP]). Dosing was on the same schedule as participants randomized to Minocin (minocycline) for Injection.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Minocin (minocycline) for Injection — Intravenous formulation of minocycline, a derivative of tetracycline
  Other Names: Minocin; Minocycline
  Arms: Minocin (minocycline) for Injection
Other: Placebo — Placebo - Normal Saline
  Arms: 0.9% Sodium Chloride Injection USP

SUMMARY:
This was a Phase 1, randomized, double-blind, placebo-controlled, single and multiple ascending dose study of the safety, tolerability, and pharmacokinetics of Minocin (minocycline) for injection in healthy adult participants.

DETAILED DESCRIPTION:
The purpose of this study was to collect safety, tolerability, and pharmacokinetic (PK) data on ascending dose regimens of Minocin (minocycline) for Injection. The safety, tolerability, and PK data was to support the compound as a potential clinical candidate in Europe and allow recommendations of dose levels to be used in future Phase 2/3 studies.

ELIGIBILITY:
Inclusion Criteria:

1. A signed informed consent form, the ability to understand the study conduct and tasks that were required for study participation, and a willingness to cooperate with all tasks, tests, and examinations as required by the protocol, whether in the research unit or after discharge, for the duration of the study
2. Male or female between 18 and 50 years of age inclusive
3. Participant had a body mass index ≥18 kilograms/square meter (kg/m^2) and ≤30 kg/m^2.
4. Participant was non-smoker or smokes up to 5 cigarettes per day (or equivalent).
5. Participant was in good health based on medical history and physical examination findings and had no clinically meaningful safety laboratory abnormalities (hematology, blood chemistry, and urinalysis) or 12-lead electrocardiogram results, as assessed by the Principal Investigator.
6. Vital signs (blood pressure, pulse, respiratory rate and temperature) measured at screening/baseline must have been within the following ranges: systolic blood pressure ≥90 to ≤150 millimeters of mercury (mm Hg), diastolic blood pressure ≥45 to ≤90 mm Hg; heart rate ≥45 to ≤90 beats per minute (taken after resting in a supine position for at least 5 minutes).
7. Expectation that intravenous access would be sufficient to allow for ease of study drug infusion, and for all protocol-required blood sampling to take place
8. Participant committed to remaining admitted in the research unit for the course of the study.
9. Female participant was surgically sterile, postmenopausal: period of amenorrhea for at least 2 years, or if of childbearing potential, agreed to abstinence or to use at least 2 acceptable methods of birth control (for example prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, barrier methods) or male partner sterilization alone, between the first dose (Day 1) and for 90 days after the completion of the study.

Exclusion Criteria:

1. Had any condition, including findings in the medical history or in pre-study assessments that constituted a risk or a contraindication for the participation in the study or completing the study
2. Positive breath test for alcohol and/or positive urine test for drugs of abuse at Screening and Day -1 Visits
3. Had a history or presence of alcohol/drug abuse within 2 years. Alcohol abuse was defined as regularly consuming >3 units/day (21 units per week for men), >2 units/day (14 units/week) for women. A unit was defined as a can of 4% beer (330 mL), approximately 190 mL of 6-7% beer (malt liquor), a glass of 40% spirits (30 mL), a glass of wine (100 mL).
4. Participant showed positive hepatitis B surface antigen, hepatitis C virus antibodies, or human immunodeficiency virus I/II antibodies and antigen tests.
5. Participant had active or ongoing candida infection.
6. Blood or plasma donation within past 2 months
7. Females who were pregnant or nursing or who had a positive pregnancy test result at the Screening Visit or Day -1 prior to dosing
8. Males who were unwilling to practice abstinence or use an acceptable method of birth control during the entire study period and for 90 days after the completion of the study (that is condom with spermicide, where locally available)
9. Presence of known raised intracranial pressure
10. Use of retinoids (for example, isotretinoin)
11. History of significant hypersensitivity or allergic reaction to any of the tetracycline class of antibiotics or the components of those antibiotics
12. Receipt of any investigational medication or investigational device during the last 30 days prior to randomization
13. Treatment with any prescription, vitamins or over-the-counter drugs, within 2 weeks or five half-lives, whichever was longer, or herbal nutritional supplements within 2 weeks of screening, with the exception of acetaminophen/paracetamol for minor headache. Participants were not allowed to receive medications for the duration of the study (except the abovementioned acetaminophen/paracetamol). Birth control or other hormone replacement were also permitted as long as it had been taken at a stable dose for at least 3 months before the Screening Visit and remained stable for the duration of the study.
14. A corrected QT interval by Fridericia >480 milliseconds
15. Calculated creatinine clearance less than 50 mL/minute (Cockcroft-Gault method) at screening or check-in (Day -1)
16. Unable or unwilling, in the judgment of the Investigator, to comply with the protocol
17. An employee of the Investigator, the study center, the sponsor or The Medicines Company with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, or a family member of the employee or the Investigator
18. Prior enrollment in any minocycline study including prior cohorts in this trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Naguib Muhsen, MD, Principal Investigator — QPS Holdings LLC
Locations (1):
- QPS, Groningen, AG, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 100 milligrams (mg) of Minocin (minocycline) for Injection on Day 1 then 100 mg every 12 hours on Days 4 to 10 and a single dose on Day 11
- Cohort 2: 200 mg of Minocin (minocycline) for Injection on Day 1 then 200 mg every 12 hours on Days 4 to 10 and a single dose on Day 11
- Cohort 3: 180 mg of Minocin (minocycline) for Injection on Day 1 then 300 mg every 12 hours on Day 4
  Due to a dosing error, participants received doses of 180 mg instead of 300 mg as planned. The cohort was discontinued on Day 5 after detection of the dosing error and replaced by Cohort 3b.
- Cohort 3b: 300 mg of Minocin (minocycline) for Injection on Day 1 then 300 mg every 12 hours on Days 4 to 10 and a single dose on Day 11
  Replacement of Cohort 3
- Cohort 4: 400 mg of Minocin (minocycline) for Injection on Day 1 then 400 mg every 12 hours on Days 4 to 7 and a single dose on Day 8
- Cohort 5: 500 mg of Minocin (minocycline) for Injection as a single dose on Day 1, 500 mg loading dose as the first dose on Day 4, 300 mg every 12 hours on Days 4 to 10 and as a single dose Day 11
- Cohort 6: 600 mg of Minocin (minocycline) for Injection as a single dose on Day 1, 600 mg loading dose as the first dose on Day 4, 300 mg every 12 hours Days 4 to 10 and as a single dose on Day 11
- Placebo: Placebo was in the form of the same 100-milliliter (mL) bags of normal saline (0.9% Sodium Chloride Injection United States Pharmacopeia [USP]). Dosing was to the same schedule as participants randomized to Minocin (minocycline) for Injection.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3b | Cohort 4 | Cohort 5 | Cohort 6 | Placebo
Started | 8 | 8 | 6 | 8 | 8 | 8 | 9 | 14
Completed | 6 | 6 | 0 (Due to an error, 180 mg given instead of 300 mg as planned. Cohort 3 was discontinued on Day 5 and replaced by Cohort 3b.) | 7 | 0 (Cohort 4 was discontinued Day 8 due to dose-limiting toxicity.) | 7 | 4 | 10
Not Completed | 2 | 2 | 6 | 1 | 8 | 1 | 5 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 1 | 6 | 1 | 4 | 0
Not completed — Sponsor Decision | 0 | 0 | 6 | 0 | 2 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: 100 mg of Minocin (minocycline) for Injection on Day 1 then 100 mg every 12 hours on Days 4 to 10 and a single dose on Day 11
- Placebo: Placebo was in the form of the same 100-mL bags of normal saline (0.9% Sodium Chloride Injection USP). Dosing was to the same schedule as participants randomized to Minocin (minocycline) for Injection.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3b | Cohort 4 | Cohort 5 | Cohort 6 | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 6 | 8 | 8 | 8 | 9 | 14 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.63 (7.76) | 31.00 (7.45) | 28.83 (9.75) | 25.00 (7.45) | 29.63 (8.72) | 25.75 (8.76) | 30.56 (12.12) | 27.43 (8.23) | 28.06 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 2 | 3 | 2 | 4 | 7 | 25
  Male | 5 | 5 | 5 | 6 | 5 | 6 | 5 | 7 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 4
  White | 8 | 7 | 6 | 8 | 7 | 6 | 7 | 14 | 63
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 8 | 8 | 6 | 8 | 8 | 8 | 9 | 14 | 69
Body Mass Index [Mean (Standard Deviation); unit: kilogram/square meter] | 23.3 (2.6) | 23.2 (2.7) | 22.5 (3.4) | 22.5 (2.4) | 22.7 (2.9) | 22.9 (2.5) | 23.4 (3.0) | 22.1 (2.8) | 22.8 (2.7)
Height [Mean (Standard Deviation); unit: centimeter] | 179.3 (9.8) | 175.8 (7.6) | 181.36 (11.2) | 178.1 (7.1) | 175.4 (9.2) | 178.0 (6.0) | 176.4 (11.0) | 178.1 (10.1) | 177.7 (8.9)
Weight [Mean (Standard Deviation); unit: kilogram] | 75.1 (10.6) | 71.7 (9.0) | 73.4 (10.1) | 71.6 (10.1) | 69.9 (11.6) | 72.6 (8.0) | 73.0 (12.7) | 70.9 (14.6) | 72.1 (11.0)

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Experiencing Treatment-emergent Adverse Events
Description: Safety and tolerability of single and multiple intravenous doses of Minocin (minocycline) for Injection assessed by number of participants with adverse events.
Time Frame: Day 1 through Day 17
Population: Safety Population: all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3b | Cohort 4 | Cohort 5 | Cohort 6 | Placebo
Number analyzed (Participants) | 8 | 8 | 6 | 8 | 8 | 8 | 9 | 14
participants
  All-Cause Mortality | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious Adverse Events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adverse Event Leading to Withdrawal from Treatment | 0 | 2 | 0 | 1 | 6 | 1 | 4 | 0
  Participants With Any Adverse Event | 6 | 8 | 4 | 8 | 8 | 8 | 9 | 12
  Participants With Any Adverse Events During Single Dose | 2 | 3 | 3 | 4 | 8 | 6 | 8 | 5
  Participants With Any Adverse Event During Multiple Doses | 6 | 7 | 3 | 8 | 7 | 8 | 8 | 12

2. Secondary Outcome: Assessment of Area Under The Concentration-time Curve From Zero Hours To The Last Measured Concentration (AUC0-t) After A Single Dose Of Minocin On Day 1
Description: Assessment of AUC0-t by cohort after a single intravenous dose of Minocin (minocycline) for Injection on Day 1 is reported as mg times hour/liter (mg*h/L).
Time Frame: Day 1 (Measurements taken at 1 [end of infusion], 2, 4, 8, 12, 18, 24, 36, 48, and 72 hours after the start of dosing)
Population: Cohort 3 PK samples were not analyzed due to early termination of the cohort. The number of participants analyzed reflects the actual number of participants with PK measurements taken at Day 1.
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3b | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 9
mg*h/L | 8.66 (1.6) | 24.0 (6.5) | 37.35 (13.9) | 59.79 (16.0) | 51.49 (20.0) | 78.98 (28.2)

3. Secondary Outcome: Assessment Of AUC0-t By Cohort After A Single Dose Of Minocin On Day 4
Description: Assessment of AUC0-t by cohort after a single dose of Minocin (minocycline) for Injection using plasma from serial blood samples on Day 4 is reported.
Time Frame: Day 4 (Measurements taken at 1 [end of infusion], 2, 4, 8, and 12 hours after the start of dosing)
Population: Cohort 3 PK samples were not analyzed due to early termination of the cohort. The number of participants analyzed reflects the actual number of participants with PK measurements taken at Day 4.
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3b | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 7 | 8 | 8 | 7 | 8 | 8
mg*h/L | 5.12 (0.9) | 11.69 (2.6) | 20.04 (7.8) | 28.54 (7.8) | 27.86 (10.0) | 42.83 (19.3)

4. Secondary Outcome: Assessment Of AUC0-t By Cohort After Multiple Doses Of Minocin On Day 11
Description: Assessment of AUC0-t by cohort after 7 days of multiple doses of Minocin (minocycline) for Injection using plasma from serial blood samples on Day 11 is reported.
Time Frame: Day 11 (Measurements taken at 1 [end of infusion], 2, 4, 8, 12, 18, 24, 36, 48, and 72 hours after the start of dosing)
Population: Cohort 3 and Cohort 4 PK samples were not taken at Day 11 due to early termination of the cohorts. The number of participants analyzed reflects the actual number of participants with PK measurements taken at Day 11.
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3b | Cohort 5 | Cohort 6
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 4
mg*h/L | 27.5 (5.5) | 80.7 (19.9) | 173.7 (100.9) | 124.1 (50.2) | 119.0 (56.3)

5. Secondary Outcome: Assessment Of Maximum Plasma Concentration (Cmax) By Cohort For A Single Dose Of Minocin On Day 1
Description: Assessment of Cmax by cohort for a single intravenous dose of Minocin (minocycline) for Injection using serial blood samples on Day 1 is reported.
Time Frame: Day 1 (Measurements taken at 1 [end of infusion], 2, 4, 8, 12, 18, 24, 36, 48, and 72 hours after the start of dosing)
Population: Cohort 3 PK samples were not analyzed due to early termination of cohort. The number of participants analyzed reflects the number of participants who had plasma PK samples taken at Day 1.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Cohort 4: 400 mg of Minocin (minocycline) for Injection on Day 1 then every 400 mg 12 hours on Days 4 to 7 and a single dose on Day 8
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3b | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
mg/L | 0.99 (0.2) | 1.89 (0.4) | 3.35 (1.2) | 4.93 (1.9) | 4.36 (0.9) | 7.03 (2.4)

6. Secondary Outcome: Assessment of Cmax by Cohort for a Single Dose of Minocin on Day 4
Description: Assessment of Cmax by cohort for a single intravenous dose of Minocin (minocycline) for Injection using serial blood samples on Day 4 is reported.
Time Frame: Day 4 (Measurements taken at 1 [end of infusion], 2, 4, 8, and 12 hours after the start of dosing)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3b | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 7 | 8 | 8 | 7 | 8 | 8
mg/L | 0.96 (0.23) | 2.05 (0.5) | 3.52 (1.6) | 4.49 (0.8) | 5.14 (1.3) | 6.51 (2.5)

7. Secondary Outcome: Assessment Of Cmax By Cohort For Multiple Doses Of Minocin On Day 11
Description: Assessment of Cmax by cohort after 7 days of twice daily dosing of Minocin (minocycline) for Injection using serial blood samples on Day 11 is reported.
Time Frame: Day 11 (Measurements taken at 1 [end of infusion], 2, 4, 8, 12, 18, 24, 36, 48, and 72 hours after the start of dosing)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3b | Cohort 5 | Cohort 6
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 4
mg/L | 1.71 (0.2) | 4.59 (1.1) | 8.91 (4.5) | 7.58 (2.4) | 6.17 (1.7)

8. Secondary Outcome: Assessment Of Apparent Terminal Elimination Half-life (T1/2) By Cohort For A Single Dose Of Minocin Using Plasma From Serial Blood Samples On Day 1
Description: Assessment of T1/2, defined by T1/2 = natural log of 2 divided by elimination constant (Kel) (T1/2), by cohort after a single intravenous dose of Minocin (minocycline) for Injection on Day 1 is reported.
Time Frame: Day 1 (Measurements taken at 1 [end of infusion], 2, 4, 8, 12, 18, 24, 36, 48, and 72 hours after the start of dosing)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Groups:
- Cohort 4: 400 mg of Minocin (minocycline) for Injection on Day 1 then 400 mg every12 hours on Days 4 to 7 and a single dose on Day 8
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3b | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 9
h | 11.05 (2.1) | 13.70 (2.3) | 16.62 (3.9) | 17.55 (2.1) | 14.44 (2.7) | 17.27 (3.6)

9. Secondary Outcome: Assessment Of T1/2 By Cohort After Multiple Doses Of Minocin Using Plasma From Serial Blood Samples On Day 11
Description: Assessment of T1/2, defined by T1/2 = natural log of 2 divided by Kel (T1/2), by cohort after 7 days of twice daily dosing of intravenous doses of Minocin (minocycline) for Injection on Day 11 is reported.
Time Frame: Day 11 (Measurements taken at 1 [end of infusion], 2, 4, 8, 12, 18, 24, 36, 48, and 72 hours after the start of dosing)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3b | Cohort 5 | Cohort 6
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 4
h | 15.89 (2.8) | 18.22 (2.4) | 19.78 (3.4) | 18.15 (1.4) | 20.19 (4.2)

10. Secondary Outcome: Assessment Of Amount Of Drug Excreted In Urine After A Single Dose Of Minocin Using Serial Urine Samples On Day 1
Description: Assessment of amount of drug excreted in urine after a single intravenous dose of Minocin (minocycline) for Injection using serial urine samples on Day 1 is reported.
Time Frame: Day 1 (Measurements collected from 0-4, 4-8, 8-12, 12-24, 24-48, and 48-72 hours after the start of dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3b | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 9
L/h | 0.37 (0.17) | 0.37 (0.04) | 0.38 (0.13) | 0.34 (0.10) | 0.40 (0.09) | 0.37 (0.13)

11. Secondary Outcome: Assessment Of Amount Of Drug Excreted In Urine After Multiple Intravenous Doses Of Minocin Using Serial Urine Samples On Day 11
Description: Assessment of amount of drug excreted in urine after 7 days of twice daily intravenous doses of Minocin (minocycline) for Injection using serial urine samples on Day 11 is reported.
Time Frame: Day 11 (Measurements collected from 0-4, 4-8, 8-12, 12-24, 24-48, and 48-72 hours after the start of dosing
Population: Cohort 3 and Cohort 4 PK samples were not taken at Day 11 at Day 11 due to early termination of the cohorts. The number of participants analyzed reflects the actual number of participants with urine samples taken at Day 11.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3b | Cohort 5 | Cohort 6
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 4
L/hr | 0.47 (0.10) | 0.35 (0.10) | 0.28 (0.09) | 0.35 (0.10) | 0.43 (0.22)

12. Secondary Outcome: Assessment Of Percent of Dose Excreted In Urine After A Single Dose Of Minocin Using Serial Urine Samples On Day 1
Description: Assessment of percent of dose excreted in urine after a single intravenous dose of Minocin (minocycline) for Injection using serial urine samples on Day 1 is reported.
Time Frame: Day 1 (Measurements collected from 0-4, 4-8, 8-12, 12-24, 24-48, and 48-72 hours after the start of dosing)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of dose
Groups:
- Cohort 5: 500 mg of Minocin (minocycline) for Injection as a single dose on Day 1, 500 mg loading dose as the first dose on Day 4, 300 mg every 12 hours Days 4 to 10 and as a single dose on Day 11
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3b | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 9
percentage of dose | 3.56 (1.54) | 4.73 (1.13) | 4.58 (0.82) | 4.98 (0.62) | 4.05 (0.50) | 4.67 (1.12)

13. Secondary Outcome: Assessment Of Percentage Of Drug Excreted In Urine After Multiple Intravenous Doses Of Minocin Using Serial Urine Samples On Day 11
Description: Assessment of percentage of drug excreted in urine after 7 days of twice daily intravenous doses of Minocin (minocycline) for Injection using serial urine samples on Day 11 is reported.
Time Frame: Day 11 (Measurements collected from 0-4, 4-8, 8-12, 12-24, 24-48, and 48-72 hours after the start of dosing
Population: Cohort 3 and Cohort 4 PK samples were not taken at Day 11 due to early termination of the cohorts. The number of participants analyzed reflects the actual number of participants with urine PK samples taken at Day 11.
Measure: Mean (Standard Deviation); unit: Percentage of dose
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3b | Cohort 5 | Cohort 6
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 4
Percentage of dose | 5.86 (0.63) | 5.80 (1.27) | 5.92 (0.72) | 6.13 (1.53) | 6.09 (1.23)

ADVERSE EVENTS:
Time Frame: All AEs occurring from the time when first dose was administered (Day 1) up to the last follow-up visit (Day 17).
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3b | Cohort 4 | Cohort 5 | Cohort 6 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/6 | 0/8 | 0/8 | 0/8 | 0/9 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/6 | 0/8 | 0/8 | 0/8 | 0/9 | 0/14
Other Adverse Events (participants affected / at risk) | 6/8 | 8/8 | 4/6 | 8/8 | 8/8 | 8/8 | 9/9 | 12/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=8) | Cohort 3 (N=6) | Cohort 3b (N=8) | Cohort 4 (N=8) | Cohort 5 (N=8) | Cohort 6 (N=9) | Placebo (N=14)
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 2 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 6 | 0 | 6 | 5 | 6 | 8 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 1 | 3 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 1
Infusion site reaction (General disorders) | 5 | 7 | 1 | 7 | 1 | 6 | 6 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 0 | 2 | 2 | 3 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 4 | 1 | 8 | 8 | 8 | 7 | 4
Headache (Nervous system disorders) | 1 | 4 | 2 | 0 | 3 | 4 | 5 | 3
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 4 | 6 | 3
Dizziness postural (Nervous system disorders) | 1 | 2 | 0 | 0 | 3 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 0
Catheter site related reaction (General disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Infusion site pain (General disorders) | 0 | 1 | 0 | 0 | 5 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeling cold (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Coordination abnormal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Substance use (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT02802631/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT02802631/SAP_001.pdf